CLINICAL TRIAL: NCT06579560
Title: Audio Vestibular Assessment in Patients with Fibromyalgia
Status: Recruiting | Type: Observational
Sponsor: Noha Osman (Other)
Responsible Party: Sponsor-Investigator, Noha Osman, Dr, Assiut University
Organization: Assiut University (Other)
Other Study IDs: 04-2023-200637
Record Dates: First submitted 2024-08-12; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Fibromyalgia
Keywords: Audiovestibular assessment, Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Audiovestibular assessment in Patients with Fibromyalgia — Audiovestibular assessment in Patients with Fibromyalgia

SUMMARY:
Fibromyalgia (FM) is a common rheumatic illness distinguished by chronic pain, fatigue, cognitive problems, and functional disability. However, the differences between men and women have not yet been comprehensively studied, especially after the development of the last 2016 American College of Rheumatology (ACR) criteria. The disease is more common and more severe in female patients according to a study on gender differences among Egyptian patients (A. Moshrif et al., 2023)

DETAILED DESCRIPTION:
Fibromyalgia (FM) is a common rheumatic illness distinguished by chronic pain, fatigue, cognitive problems, and functional disability. However, the differences between men and women have not yet been comprehensively studied, especially after the development of the last 2016 American College of Rheumatology (ACR) criteria. The disease is more common and more severe in female patients according to a study on gender differences among Egyptian patients (A. Moshrif et al., 2023) (FM) is a non-inflammatory chronic disease, characterized by widespread musculoskeletal pain (Tuncer et al., 2021). The etiology is still unknown and (FM) is often misdiagnosed (Tuncer et al., 2021).The estimated prevalence in the general population is between 2 and 11% (Hulens et al., 2023). Although the underling Pathological mechanisms controlling the (FM) have not been determined, neuroendocrine, genetic or molecular factors can be involved (Zeigelboim & Moreira, 2011).(FM) affects females between the ages of 25 to 65 years old, although it can be seen in all ages and in both sexes (Fitzcharles & Yunus, 2012), It's more common in females than in males (Müller et al., 2007).

The main symptoms of (FM) include, muscle pain, muscle spasms, insomnia, fatigue, tension, abdominal pain, facial tenderness, sensitivity to noise and bright lights, and central nervous system abnormalities. Various neurological symptoms such as tinnitus, ear fullness, vertigo, and dizziness may also be associated, regardless of the disease severity (Koca et al., 2018) Many patients with FM were reported to have dizziness which may attributed to hypotension and autonomic nervous system (ANS) dysfunction, in this study we want to explore if dizziness and imbalance occur due to these factors only or due to a direct effect of (FM) on the vestibular system (Kanjwal et al., 2010) (Mohamed et al., 2021).

ELIGIBILITY:
1. Inclusion criteria: - Age: 15-50 years.

   * Sex: Male & Female.
   * Patients with fulfilling the criteria for the diagnosis of FM
2. Exclusion criteria: Patients not fulfilling the criteria for the diagnosis of FM.

   * Other causes of SNHL as Meniere's disease.
   * Other causes of Conductive hearing loss (CHL) as chronic suppurative otitis media CSOM.
   * Other causes of collagen and connective tissue diseases.
   * Abnormal EMG.
   * Abnormal radiological studies of the brain.
   * Patients are receiving of ototoxic drugs.

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients diagnosed with Fibromyalgia recruited from the Rheumatology and Rehabilitation Department at Al-Azhar University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 4 (Estimated)
Dates: Start 2023-04-16 (Actual); Primary Completion 2025-04-16 (Estimated); Study Completion 2025-04-16 (Estimated)

PRIMARY OUTCOMES:
Hearing Sensitivity | 2 years
  Measurement of hearing sensitivity using pure tone audiometry. The outcome will be expressed as hearing thresholds in decibels (dB) at various frequencies (e.g., 250 Hz, 500 Hz, 1000 Hz, 2000 Hz, 4000 Hz).
  [Unit of Measure: Decibels (dB)]

CONTACTS AND LOCATIONS:
Overall Officials: Enass S. Mohamed, Professor, Study Chair — Assiut University; Abdelhafeez M. Moshrif, Professor, Study Chair — Assiut University; Mohamed A. Elmoursy, Professor, Study Chair — Assiut University
Locations (1):
- Faculty of Medicine - Assiut University, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No